CLINICAL TRIAL: NCT00134355
Title: Phase II Evaluation of PTK787, an Oral Vascular Endothelial Growth Factor Inhibitor, in Patients With Non-Metastatic Androgen Independent Prostate Cancer
Brief Title: Study of PTK787 in the Treatment of Patients With Non-Metastatic Androgen Independent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2005.014
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Prostate Cancer
Keywords: antiangiogenesis therapy; vatalanib
MeSH Terms: conditions — Prostatic Neoplasms | interventions — vatalanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PTK787 (Experimental): PTK787:
  250 mg orally twice daily x 2 wks, then 250 mg orally am, 500 mg orally pm x 1 wk, then 500 mg orally twice daily
  Interventions: Drug: PTK787

INTERVENTIONS:
Drug: PTK787

SUMMARY:
The purpose of this study is to evaluate PTK787/ZK 222584, a drug that blocks new blood vessel growth, in the treatment of patients with non-metastatic androgen independent prostate cancer. This study will assess the safety and tolerability of PTK787/ZK 222584, and evaluate serum vascular endothelial growth factor (VEGF) levels.

DETAILED DESCRIPTION:
This is an open-label, phase II trial of PTK787/ZK 222584. Patients will receive 750 mg daily for one week, 1000 mg daily for the second week, and then 1250 mg per day thereafter.

Response Assessment: In the absence of toxicity or clinical progression, patients will remain in the study until their PSA (Prostate-specific Antigen) has doubled from pretreatment baseline.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of prostate cancer
* No evidence of metastatic disease
* PSA-only progression despite androgen depravation therapy and antiandrogen withdrawal
* Patients must maintain castrate levels of testosterone (<50ng/mL) or continue on LHRH ( Luteinizing Hormone-releasing Hormone) analog therapy.
* ECOG (Eastern Cooperative Oncology Group) performance status of 0-2 (A measure of quality of life where 0 represents asymptomatic and 5 represents death)
* No prior anti-VEGF therapy is allowed
* No investigational or commercial agents or therapies other than LHRH agonists/antagonists may be administered concurrently with intent to treat the patient's malignancy
* Age greater than or equal to 18 years
* Life expectancy greater than 6 months
* Normal organ and marrow function obtained within 14 days prior to registration
* Must use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Patients may continue on a daily multivitamin, but all other herbal or alternative food supplements must be discontinued before registration.
* Patients must be on stable doses of bisphosphonates which have been started no less than 6 weeks prior to protocol therapy.
* Uncontrolled incurrent illness
* Patients with a "currently active" second malignancy are not eligible.
* Major surgery less than or equal to 4 weeks prior to randomization
* Prior chemotherapy less than or equal to 3 weeks prior to registration
* Prior biologic or immunotherapy less than or equal to 2 weeks prior to registration
* Prior investigational drugs of any kind less than or equal to 4 weeks prior to registration
* Patients who have had full field radiotherapy less than or equal to 4 weeks or limited field radiotherapy equal or less than 2 weeks prior to registration.
* Patients must not be on nonsteroidal antiandrogen blockade.
* Patients must have no evidence of disease on bone scan or computed tomography (CT) scan of the abdomen/pelvis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-07; Primary Completion 2006-11 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Time To Progression (TTP) in Weeks | 12 Months

SECONDARY OUTCOMES:
Number of Toxicities in Patients Treated with PTK787 | 30 Days After Last Dose
Overall Survival | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen W. Beekman, MD, Principal Investigator — The University of Michigan Comprehensive Cancer Center